CLINICAL TRIAL: NCT05746169
Title: DREAM: Discovering Cancer Risks From Environmental Contaminants And Maternal/Child Health
Brief Title: Discovering Cancer Risks From Environmental Contaminants and Maternal/Child Health
Status: Terminated | Type: Observational
Why Stopped: Collaborating funding sponsor decision
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); California Office of Environmental Health Hazard Assessment (OEHHA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21621; NCI-2022-10633 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); UG3CA265845 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Cancer Risk; Environmental Cancer Risk; Maternal-Child Cancer Risk; Environmental Contaminants
MeSH Terms: conditions — Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal urine will be collected at 2nd trimester, delivery, and 4-year visit.
  * Maternal blood will be collected at 2nd trimester, delivery, and 4-year visit. Self-collected maternal blood will be collected via finger stick.
  * Maternal hair and nail samples will be collected at 2nd trimester , 2.5-year assessment, and 4-year assessment. Toenail samples will be collected with standard, stainless steel toenail clippers.
  * Umbilical cord blood samples will be collected at time of delivery.
  * Child hair and nail samples will be collected at two timepoints: 2.5-year follow-up assessment and 4-year clinic visit.
  * Child urine will be collected from children at the 4-year clinic visit.
  * Child saliva will be collected from saliva samples from children at the 4-year clinic visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their children: The DREAM cohort will recruit from University of California, San Francisco (UCSF) Mission Bay, Zuckerberg San Francisco General Hospital, and Fresno Community Medical Center locations to enroll an economically, geographically, ethnically and racially diverse cohort of pregnant women and their children for long term follow-up.
  Interventions: Other: Health Questionnaires; Other: Specimen sample collection

INTERVENTIONS:
Other: Health Questionnaires — A questionnaire with content developed and tested in the investigator's previous reproductive and cancer epidemiology studies as part of the NIH Environmental Influences on Child Health Outcomes (ECHO) consortium will be used to collect information on primary established and hypothesized risk factors for cancer and additional covariates.
Other: Specimen sample collection — Collection of blood, urine, nails, hair, and saliva samples will be obtained during the participant encounters.
  Other Names: Biospecimen sample collection; Specimen collection

SUMMARY:
The DREAM Cohort is a longitudinal observational study developed to enhance our understanding of how multiple exposures to environmental chemicals and pollutants across a diverse population of pregnant women and their offspring are linked to cancer risks. Because pregnancy induces multiple maternal hormonal and physiological changes that can increase cancer susceptibility to environmental chemical exposures, this study will focus on pregnancy as a period of particular vulnerability to toxic agents.

DETAILED DESCRIPTION:
The environmental exposures will focus on two major components: Consumer product related chemicals (including per- and polyfluoroalkyl substances (PFAS), phthalates and plasticizers, phenolic compounds, pesticides, and aromatic amines) measured via biomonitoring and prioritized based on widespread public exposure; and environmental pollutants in air and water, evaluated via geographic information system analyses of participants' residential histories.

The study team will collect questionnaire data and biospecimen samples starting at the second trimester of pregnancy up until the child reaches four years of age. A Cohort Ambassador Program will also be established to invite participants across our three sites to provide continuous feedback which will be integrated into the research priorities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, over the age of 18 years.
* English or Spanish-speaking.
* Children born of participants enrolled during pregnancy will be enrolled in the DREAM cohort.
* Inclusion criterion for the DREAM Cohort Ambassador Program is limited to research participants in the DREAM Cohort.

Exclusion Criteria:

* Women under the age of 18.
* Women expecting the birth of multiples (twins, triplets, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their children
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Assessment of levels of consumer product-related chemicals | Up to 4 years
  Consumer product related chemicals measured via biomonitoring of polyfluoroalkyl substances (PFAS), phthalates and other plasticizers, phenolic compounds, pesticides, and aromatic amines will be assessed.
Evaluation of endocrine system disruptions | Up to 4 years
  Exposures to environmental chemicals that disrupt endocrine and related biological systems during pregnancy which may predispose women and children to cancer will be evaluated.
Assessment of Inflammation/Immune modulation | Up to 4 years
  Measures of peripheral whole blood using a standard laboratory procedure for Complete Blood Count (CBC) panel will be calculated to assess shifts in immune cell profiles indicative of inflammation and immune modulation.
Impact of geographical environmental pollutants | Up to 4 years
  The environmental pollutants found in air and water, as well as pesticide use, will be evaluated via geographic information system analyses of participants' residential history.
Frequency of oxidative stress biomarkers | Up to 4 years
  Oxidative Stress/DNA damage will be measured by seven oxidative stress biomarkers which reflect oxidative damage to DNA will be measured to determine overall assessment of oxidative damage to DNA: proteins and lipids (OSBs): (o,o -dityrosine (diY), 8-hydroxy-2 -deoxyguanosine (8-OHdG), malondialdehyde (MDA), and four F2-isoprostane isomers (i.e., 8-isoprostaglandinF2α [8-PGF2α], 11β-prostaglandinF2α [11-PGF2α], 15(R)-prostaglandinF2α [15-PGF2α], and 8-iso,15(R)-prostaglandinF2α [8,15-PGF2α]) in maternal urine.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Reynolds, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Berkeley, Berkeley, California
  - Fresno Community Regional Medical Center, Fresno, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No